CLINICAL TRIAL: NCT04978376
Title: Time Restricted Eating With Physical Activity for Weight Management
Brief Title: TRE With Physical Activity for Weight Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Kelsey Nicole Dipman Gabel, Clinical Assistant Professor and Postdoc, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-0575
Record Dates: First submitted 2021-07-22; First posted 2021-07-27 (Actual); Results first posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-09

CONDITIONS: Pre Diabetes; Overweight and Obesity
Keywords: Intermittent Fasting
MeSH Terms: conditions — Glucose Intolerance; Overweight; Obesity; Intermittent Fasting | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Time restricted eating (Experimental): ad-libitum eating between 12:00-20:00
  Interventions: Behavioral: Time restricted eating
- TRE with endurance training (Experimental): ad-libitum eating between 12:00-20:00 with 3-5 days of supervised endurance exercise per week
  Interventions: Behavioral: Time restricted eating
- TRE with resistance training (Experimental): ad-libitum eating between 12:00-20:00 with 3-5 days of supervised resistance training per week
  Interventions: Behavioral: Time restricted eating
- Control (No Intervention): no change in diet or physical activity

INTERVENTIONS:
Behavioral: Time restricted eating — We will compare the effects of time restricted eating alone and combined with resistance exercise of endurance exercise versus a no intervention control group.
  Other Names: resistance training; endurance exercise
  Arms: TRE with endurance training; TRE with resistance training; Time restricted eating

SUMMARY:
Approximately 24 million older adults have prediabetes. Obesity, age related decreases in lean mass and increases in fat mass, and sedentary lifestyle have been associated with functional and cognitive decline in older adults. Innovative lifestyle strategies to treat obesity and pre-diabetes are critically needed. The proposed research will demonstrate that time restricted eating combined with resistance training is an effective non-pharmacological therapy to help obese prediabetic individuals reduce body fat, maintain lean mass, prevent progression of prediabetes to diabetes, and improve cognition.

DETAILED DESCRIPTION:
Obesity, age related decreases in lean mass and increases in fat mass, and sedentary lifestyle have been associated with functional and cognitive decline in older adults. It is expected that the proportion of the population of over 65 will continue to increase as will the number of older adults with pre-diabetes. Treatment of pre-diabetes and improved functionality and cognition in older adults include maintaining a healthy weight and regular exercise. While daily calorie restriction is the most common prescription for weight loss, intermittent fasting is an alternative to daily calorie restriction producing significant weight loss. Currently, the most popular form of intermittent fasting is time restricted eating (TRE). TRE typically involves confining the eating window to 6-10 h and fasting for the remaining hours of the day. During the eating window, individuals are not required to count calories or monitor food intake in any way. Current TRE data shows promising results for diet alone including natural calorie restriction, weight loss, decreased blood pressure and increased insulin sensitivity all while maintaining a high adherence. To our knowledge, TRE combined with resistance training (RT) or endurance training (EN)has only been examined in lean resistance trained young adults, never in older adults or adults with overweight or obesity. Hypothesis: The present proposal will test the following hypothesis: (1) Both combination groups will lose significantly more weight than TRE alone or the control. The TRE + RT group will significantly decrease fat mass and increase lean mass more than the TRE + EN, TRE alone or control group. The TRE + RT will lose the same amount of body weight but maintain more lean mass than the TRE+EN group; (2a) The TRE+RT group will experience greater improvements in insulin sensitivity, insulin resistance, HbA1c and other metabolic disease variables (fasting insulin, triglycerides, LDL cholesterol, and blood pressure) versus the TRE+EN group after the 8-week trial due to reductions in body weight and greater retention of lean mass; (2b) TRE combined with both EN and RT will be safe in older adults with no significant intervention related adverse events; (3) TRE combined with both EN and RT will improve attention and executive function and working memory in the physical activity groups more than diet alone or the control group. Methods: To test these objectives, a 10-week parallel-arm pilot trial will be implemented. Older adults with overweight or obesity and pre-diabetes will be assigned to one of four groups: (1) TRE group, ad-libitum eating between 12:00-20:00 (n=50) (2) TRE + EN ad-libitum eating between 12:00-20:00 with 3-5 days of supervised endurance exercise per week (n=50) (3)TRE + RT group, ad-libitum eating between 12:00-20:00 with 3-5 days of supervised resistance training per week (n=50) or (4) Control group, no change in diet or physical activity (n=50). Significance: If the aims of this application are achieved, this study will be the first to show that TRE with physical activity is safe in older adults and can be implemented as an alternative to traditional dieting (i.e. daily calorie restriction) for weight management and lean mass retention. This study will also show that TRE can be used as an effective non-pharmacological therapy to improve insulin sensitivity, decrease metabolic risk factors, and improve cognition in older individuals with obesity and pre-diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 to 70 years old
* BMI between 25 and 50 kg/m2
* Pre-diabetic or insulin resistant (fasting glucose: 100-125 mg/dl, HBA1c 5.7%-6.4%, or HOMA-IR >2.5)
* Sedentary or lightly active 24
* Are post menopausal (absence of menstrual cycle for 1 year)

Exclusion Criteria:

* Diabetic (fasting glucose: >126 mg/dl or HBA1c >6.5%)
* Have a history of eating disorders (anorexia, bulimia, or binge eating disorder)
* Have uncontrolled hypertension, any other cardiovascular disease, or history of aneurysm
* History of alcohol dependance (score >20 from Alcohol and Health Questionnaire)25
* Are not weight stable for 3 months prior to the beginning of study (weight gain or loss > 4 kg)
* Are not able to keep a food diary or activity log for 7 consecutive days during screening
* Are taking drugs that influence study outcomes (weight loss, glucose-lowering medications)
* Are premenopausal, perimenopausal or have an irregular menstrual cycle (menses that does not appear every 27-32 days)
* Mobility disability (unable to exercise for 40-60 minutes 3-5 days/week)
* Diagnosed comorbidities including systemic diseases (Parkinson's cirrhosis, renal disease or systemic rheumatic conditions), cancer, or cognitive impairment
* Are night shift workers
* Are smokers

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelsey Gabel, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Time Restricted Eating | TRE With Endurance Training | TRE With Resistance Training | Control
Started | 4 | 4 | 5 | 4
Completed | 4 | 4 | 5 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Time Restricted Eating | TRE With Endurance Training | TRE With Resistance Training | Control | Total
Number analyzed (Participants) | 4 | 4 | 5 | 4 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 5 | 4 | 15
  >=65 years | 1 | 1 | 0 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (4) | 61 (6) | 57 (6) | 52 (5) | 57 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 5 | 4 | 15
  Male | 1 | 1 | 0 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 4 | 4 | 5 | 2 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 5 | 2 | 15
  White | 0 | 0 | 0 | 2 | 2
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 5 | 4 | 17
BMI [Mean (Standard Deviation); unit: kg/m^2] | 36 (4) | 34 (3) | 36 (4) | 35 (5) | 35 (4)
Weight [Mean (Standard Deviation); unit: kilograms] | 97 (10) | 98 (20) | 97 (13) | 89 (16) | 95 (15)

OUTCOME MEASURES:

1. Primary Outcome: Body Weight Changes Between Week 1 to Week 10
Description: Body weight assessed to the nearest 0.25 kg every week without shoes and in light clothing using a balance beam scale (HealthOMeter, Boca Raton, FL).
Time Frame: Change from week 1 to week 10
Measure: Mean (Standard Error); unit: Percent body weight loss
Arm/Group | Time Restricted Eating | TRE With Endurance Training | TRE With Resistance Training | Control
Number analyzed (Participants) | 4 | 4 | 4 | 4
Percent body weight loss | -2.1 (.8) | -4.2 (.8) | -1.3 (1.1) | .1 (.5)

2. Secondary Outcome: Body Composition Changes From Week 1 to Week 10
Description: Change in lean mass from week 1 to week 10 by DEXA
Time Frame: Change from week 1 to week 10
Measure: Mean (Standard Error); unit: percent lean mass change
Arm/Group | Time Restricted Eating | TRE With Endurance Training | TRE With Resistance Training | Control
Number analyzed (Participants) | 4 | 4 | 4 | 4
percent lean mass change | -3.5 (.9) | -1.4 (.8) | .7 (.9) | -.3 (5.1)

3. Secondary Outcome: Change in Insulin From Week 1 to Week 10
Description: insulin will be measured by enzymatic kit (uIU/ml)^4
Time Frame: Change from week 1 to week 10
Population: t-test
Measure: Mean (Standard Error); unit: (uIU/ml)^4
Arm/Group | Time Restricted Eating | TRE With Endurance Training | TRE With Resistance Training | Control
Number analyzed (Participants) | 4 | 4 | 5 | 4
(uIU/ml)^4 | -.9 (.1) | .6 (.7) | .3 (2.5) | 2 (1.3)

4. Secondary Outcome: Glucose
Description: measured by enzymatic kit (mg/dl)
Time Frame: Change from week 1 to week 10
Population: t-test
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Time Restricted Eating | TRE With Endurance Training | TRE With Resistance Training | Control
Number analyzed (Participants) | 4 | 4 | 5 | 4
mg/dl | -.5 (2.2) | 1.5 (10.5) | -5 (1.8) | 1.7 (8.8)

ADVERSE EVENTS:
Time Frame: 10 weeks
Description: Time restricted eating and increases in physical activity only hold minimal risk, however serious adverse events and all cause mortality were monitored per the OSP and the OVCR.
Arm/Group | Time Restricted Eating | TRE With Endurance Training | TRE With Resistance Training | Control
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/5 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/76/NCT04978376/Prot_SAP_000.pdf